CLINICAL TRIAL: NCT06547307
Title: Effects of Caffeine, CYP1A2 and ADORA2A Genotypes on Cycling Endurance Performance.
Brief Title: CYP1A2 and ADORA2A Genotypes and Endurance Performance.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Masaryk University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: MasarykU
Record Dates: First submitted 2024-08-01; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: endurance; genotype; caffeine; ergogenic effect
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Caffeine 2 mg (Active Comparator): To compare exercise performance of 2 or 4 mg of caffeine per kilogram of body weight to placebo within subjects. Subjects will perform one exercise test (10 km cycling time trial).
  Interventions: Dietary Supplement: Caffeine 2 mg
- Caffeine 4 mg (Active Comparator): To compare exercise performance of 2 or 4 mg of caffeine per kilogram of body weight to placebo within subjects. Subjects will perform one exercise test (10 km cycling time trial).
  Interventions: Dietary Supplement: Caffeine 4 mg
- Placebo (Placebo Comparator): To compare exercise performance of 2 or 4 mg of caffeine per kilogram of body weight to placebo within subjects. Subjects will perform one exercise test (10 km cycling time trial).
  Interventions: Dietary Supplement: Caffeine 0 mg

INTERVENTIONS:
Dietary Supplement: Caffeine 2 mg — To compare exercise performance of 2 or 4 mg of caffeine per kilogram of body weight to placebo within subjects.
  Arms: Caffeine 2 mg
Dietary Supplement: Caffeine 4 mg — To compare exercise performance of 2 or 4 mg of caffeine per kilogram of body weight to placebo within subjects.
  Arms: Caffeine 4 mg
Dietary Supplement: Caffeine 0 mg — To compare exercise performance of 2 or 4 mg of caffeine per kilogram of body weight to placebo within subjects.
  Arms: Placebo

SUMMARY:
The aim of this randomized, double-blind, placebo-controlled experiment will be to assess the potential effect of the selected gene polymorphism (CYP1A2, ADORA2A) on performance after caffeine ingestion.

DETAILED DESCRIPTION:
This randomized, double-blinded, placebo-controlled, within-subjects counter-measured study design will include 60 males and females that fall between the given age range (18-35 years).

Participants will complete five visits (~90-120 min each, 2 visits during the first week,3 visit during week 2-4) in the Laboratory at Faculty of Sports Studies of Masaryk University. All testing will take place Monday to Friday during morning hours (7-12) to minimize potential diurnal effect on sports performance. Participants will be instructed to maintain their regular diet (pre-testing meals will be replicated for all visits) and sleeping habits, avoid strenuous activity 48 hours before each visit, and abstain from caffeine one week prior to the first visit and for the duration of the data collection (4 weeks).

Sample size calculations We estimated sample size using G*Power 3.1 (Version 3.1.9.4). Effect size = 0.25, the trial would be powered to detect small but still physiologically important effect.

Alpha error = 0.025 Power (1-Beta probability) = 0.8 Number of groups = 6 - number of stratification required for genotype subgroup analysis number of measurements = 3 Sample size = based on calculation, 60 participants are required

Recruitment

Recruitment will be carried out at Masaryk University by flyers. Recruitment will also take place online through sharing on the website and social networks of the Faculty of Sports Studies of Masaryk University.

Parameters of Assessment

Physiological data will be collected by a Ph.D.-level exercise physiologist and two doctoral students.

Height will be measured to the nearest 0.1 cm using a wall-mounted stadiometer, and body weight will be measured to the nearest 0.1 kg using a digital scale with participants wearing light clothing without shoes.

Body weight value will be measured on each visit and will be used to determine 2 and 4 mg per kilogram of body mass dosages for caffeine treatments (plus a placebo dose) that will be ingested in random order (derived by research assistant and blinded to all investigators) during visits 2, 3 and 4, over the following three weeks.

Body composition will be assessed by dual-energy x-ray absorptiometry (DXA; Horizon A, Hologic Inc. Marlborough, MA) during the first week of the study.

Exercise Tests

VO2max test

Each participant will initially perform an incremental exercise test. That test will assess Vo2max and maximal workload (Wmax), which is necessary for subsequent settings. Respiratory parameters will be measured breath-by-breath using a CORTEX METALYZER 3B. Wmax will be calculated using the following equation:

Wmax= Wfinal + (t/T) x Winc. Where Wfinal is the power output of the final completed stage, t is the time achieved in the final uncompleted stage (s), T is the duration of each stage (s) and Winc is the workload increment.

Time trial

The ergometer will be set to linear mode (workload increases as the pedalling rate increases). Each participant will perform a warm-up at 1 W/kg for 5 minutes. After the warm-up participants will be instructed to complete 10 km trial as quickly as possible (with no temporal, verbal, or physiological feedback). The primary variable measured will be the time to completion of the 10 km TT. The ergometer will be set to linear mode using the following formula:

W = L x (rpm)2, where rpm is the pedalling rate and L is a linear factor dependent on the participant's Wmax. To ensure consistency across participants, the resistance on the pedals during the TT will be set so that the participants would achieve 60 % of their power output at 80 rpm using the following equation:

L = (0.60 x Wmax)/6400

A familiarization time trial will occur during the first week of a study.

Rate of perceived exertion

During the time trial protocol, information about the rate of perceived exertion will be collected. Participants will be shown a Borgs scale of Perceived Exertion to assess the subject's fatigue, This will be performed twice during the time trial protocol (5th and 9th km)

Genotyping

Buccal mucosa smears will be collected during the first week of the study. Investigators will examine known genetic variations (CYP1a2 (rs 762551), ADORA2A (rs 5451876)) that are associated with caffeine metabolism and response, to determine if these genes affect response to exercise after subjects ingest caffeine.

Caffeine intake questionnaire

Investigators will use a Caffeine intake questionnaire - revised (CCQ-R) to determine habitual caffeine intake in the week before the study starts and then each week to discover whether the participants comply with the restriction regarding caffeine, or whether they have started consuming, for example, more chocolate

Training status

At the beginning of the study, participants with one of the study investigators will complete Training and Performance Caliber: A Participant Classification Framework, based on the study by McKay et al., 2021 to determine the training status of each individual.

Statistical analysis

The statistical analysis will be carried out using IBM SPSS software. Descriptive data will be reported (VO2max/peak, body height, body weight, %body fat, lean body mass, habitual caffeine intake, training status. A t-test will determine the comparison between genotypes. Potential differences between 10 km TT will be assessed by an ANOVA with treatment as a within-participants factor and genotype as a between-participants factor.if the distribution of the data will not be normal, we will apply non-parametric equivalent of the test

Experimental procedure

Week 1

There will be three visits to the laboratories of the Faculty of Sports Studies at Masaryk University (FSpS MU):

i. Participants will undergo body composition measurement (DXA) and a cheek swab for assessing selected gene variants. Data about height, weight and age will be collected (Day 1: approximate duration of visit to FSpS MU 60-90 minutes).

ii. Participants will undergo maximal load testing using a cycling ergometer test and critical power testing using a cycling ergometer test (Day 2: approximate duration of visit to FSpS MU 90 minutes).

iii. Participants will practice a 10-km time trial on the cycling ergometer (Day 3: approximate duration of visit to FSpS MU 60 minutes).

Weeks 2, 3, 4

Participants will undergo a 10-km time trial on the cycling ergometer. After arrival participants will be randomly assigned to one of the three conditions. They will always ingest same amount of the identical capsules (with same colour, size). After 50 minutes after the capsule ingestion, participants will start the warm-up and 60 minutes after the ingestion the TT will start. This procedure will be identical for all experimental week (2, 3 and 4). Participants may drink water ad libitum throughout the exercise test.

ELIGIBILITY:
Inclusion Criteria:

* healthy person
* any training status
* within age limits
* without contraindications to perform the test on a bicycle trainer
* No contraindications to caffeine intake

Exclusion Criteria:

* Pregnancy
* Breast feeding
* Cardiovascular disease
* Hypertension
* Liver disease in the previous two months
* Taking drugs that can affect liver function
* Illness in the period of 14 days before the start of the research
* Use of caffeine during research

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Efficacy of caffeine to improve endurance performance (time to complete 10 km trial) | 2 Hours
  To determine if caffeine intake improves endurance performance compared to placebo. Efficacy of caffeine doses (2 mg/kg and 4 mg/kg) to shorten the time needed to complete the 10 km time trial.

SECONDARY OUTCOMES:
Caffeine ingestion and genotype interaction | 1 day
  To determine if different variants of selected genes affect the potential ergogenic effect of caffeine. A buccal mucosa smear will be taken to identify variants of CYP1A2 and ADORA2A genes to determine which genes/variants are associated with improvement in time trial performance after caffeine ingestion.

CONTACTS AND LOCATIONS:
Overall Officials: Lucie Lipková, Principal Investigator — Masaryk University
Locations (1):
- Masaryk University, Brno, Czechia